CLINICAL TRIAL: NCT05910788
Title: High-Flow Nasal Catheter (HFNC) Compared With Conventional Oxygenation During the Perioperative Period of Patients Undergoing Thoracic Surgery.
Brief Title: High-Flow Nasal Catheter (HFNC) Compared With Conventional Oxygenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Desire Tarso Maioli, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: U1111-1292-9259
Record Dates: First submitted 2023-05-29; First posted 2023-06-20 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Thoracic Surgery
Keywords: Thoracic surgery; High flow nasal cannula; Pulmonary complications

STUDY DESIGN:
Intervention Model Description: Main goal
  * To evaluate the incidence of in-hospital pulmonary complications in 30 days in patients submitted to the use of HFNC in the perioperative period of patients undergoing thoracic surgery,
  * To evaluate in-hospital postoperative mortality within 30 days.
  intubation)
  Secondary objectives
  * Assess the incidence of hypoxemia during orotracheal intubation/ extubation
  * Assess the incidence of immediate complications after intubation/ extubation(desaturation, failure of intubation/ extubation)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC (Active Comparator): The intervention group will receive HFNC therapy at induction of anesthesia. The intervention group will receive oxygen by 100% HFNC with a flow of 40 L.min-1 being increased to 70 L.min-1 during the period of apnea. A rapid sequence of orotracheal intubation will be performed, considering the time of apnea the moment of disappearance of the capnography line until the first ventilation after tube placement.
  Interventions: Device: high flow nasal cannula
- Convencional oxygen therapy (No Intervention): Control group will receive conventional oxygen therapy by mask facial, with 100% oxygen and flow of 10 L.min-1.After surgery, patients who are extubated in the operating room or in theintensive care unit, will remain in the control and intervention groups and will receive therapy for conventional oxygen or HFNC, respectively.

INTERVENTIONS:
Device: high flow nasal cannula — The purpose of this intervention is clarify the benefit with the perioperative use of HFNC, in thoracic surgeries, from intubation to the postoperative period, evaluating mortality and in-hospital complications.
  is to clarify whether there is benefit from the perioperative use of HFNC, in thoracic surgeries, from intubation to the postoperative period, evaluating mortality and in-hospital complications.
  Arms: HFNC

SUMMARY:
The purpose of this study, is to clarify whether there is benefit from the perioperative use of HFNC in thoracic surgeries, from intubation to the postoperative period, evaluating hipoxemia during orotracheal intubation, immediate complications after intubation, mortality and in-hospital complications.

DETAILED DESCRIPTION:
High-flow Nasal Catheter (HFNC) compared to oxygenation conventional during the perioperative period of patients undergoing thoracic surgery The increase in surgeries performed worldwide, with today an estimate of more than 300 million surgeries/year, makes us increasingly need knowledge and strategies to improve perioperative care. Complications in this period are responsible for an increase in morbidity and mortality of patients, reducing the effectiveness of the surgical treatment, mainly in developing countries. The use of a nasal cannula high-flow (HFNC) oxygen during the perioperative period offers a promising technique to improve the lung function of these patients, enabling better outcomes.

The purpose of this study, therefore, is to clarify whether there is benefit from the perioperative use of HFNC, in thoracic surgeries, from intubation to the postoperative period, evaluating mortality and in-hospital complications.

Primary and secondary objectives

Main goal

* To evaluate the incidence of in-hospital pulmonary complications in 30 days in participants submitted to the use of HFNC in the perioperative period of participants undergoing thoracic surgery, when compared to the use of conventional oxygen therapy.
* To evaluate in-hospital postoperative mortality within 30 days.

Secondary objectives

* Assess the incidence of hypoxemia during orotracheal intubation and extubation
* Assess the incidence of immediate complications after intubation and extubation (desaturation, failure of intubation/ extubation)

It will be a randomized, non-blinded, single-center clinical trial. Participants (older than 18 years old) who undergo thoracic surgery and who are at surgical risk for postoperative complications with ARISCAT > 26 (risk score for pulmonary complications) will be allocated consecutively and randomized to participate in the intervention group or control, receiving written informed consent to the study and interventions. The study will be carried out at Hospital Tacchini, from July 2023 to June 2024.

Control group will receive conventional oxygen therapy, and the intervention group will receive HFNC therapy at induction of anesthesia and postoperatively, after extubation.

Oxygenation will be performed, according to the randomization, in the control group, by mask facial, with 100% oxygen and flow of 10 L.min-1. The intervention group will receive oxygenby 100% HFNC with a flow of 40 L.min-1 being increased to 70 L.min-1 during the periodof apnea.

A rapid sequence of orotracheal intubation will be performed, considering the time of apnea the moment of disappearance of the capnography line until the first ventilation after tube placement. Difficulties and complications in carrying out this step will be described. A oxygen saturation will be measured before the start of pre-oxygenation and will be considered hypoxemia, any measurement below 90% saturation, during the initiation of the rapid sequence intubation up to 5 minutes after it, in both groups. All participants will be intubated according to current orotracheal intubation guidelines. After surgery, participants who are extubated in the operating room or in the intensive care unit, will remain in the control and intervention groups and will receive therapy for conventional oxygen or HFNC, respectively. The fraction of inspired oxygen (FiO2) will be titrated until pulse oximetry is above 95%, which is also reduced to the level minimum, to achieve this objective. In the control group, oxygen will be offered through a nasal catheter or face mask and those in the intervention group will receive oxygen through HFNC with flows adjusted between 30 and 50 L.min-1, depending on the respiratory rate (less than 16) and the patient comfort.

Data and statistics analysis strategy The data, after being collected, will be expressed as mean and standard deviation or absolute frequency and relative. Data normality will be tested by the Kolmogorov-Smirnov test. The difference Significant difference between groups will be analyzed using Student's t test for data for parametric data and for non-parametric data the Wilcoxon test will be used. The program used will be the Statistical Package for the Social Sciences, version 20 (SPSS Inc., Chicago, IL,USA) and the significance level adopted will be p<0.05.

Calculation and/or justification of the sample size According to the literature, patients undergoing thoracic surgery may present severe complications such as postoperative hypoxemia in up to 30% of cases, after extubation. Based on the literature review, the sample calculation should be 45 patients for each group. For the sample calculation, we considered the value of β of 20% and α of 5%.

. Using a effect size (calculated from the article data) of 0.6, a statistical power of 80% and a significance level of p<0.05 (or 5%), the investigators obtained as a result the n of 90 volunteers per group (final sample, excluding possible losses). The G*Power program version 3.1.9.2 for Windows (Franz Faul, University Kiel, Germany) was used to perform the calculation.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age who will undergo elective thoracic surgery and who have an ARISCAT score > 26.

Exclusion Criteria:

* Patients who need urgent/emergency surgery, pregnant women, who do not have an ARISCAT score > 26 and those who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Complications | 30 days
  To evaluate the incidence of in-hospital pulmonary complications in 30 days in patients submitted to the use of HFNC in the perioperative period of patients undergoing thoracic surgery, when compared to the use of conventional oxygen therapy. extubation
Mortality | 30 days
  To evaluate in-hospital postoperative mortality within 30 days.

SECONDARY OUTCOMES:
Incidence of hipoxemia | 5 minuts
  - Assess the incidence of hypoxemia during orotracheal intubation and extubation.
Complications after intubation and extubation | 5 minuts
  Assess the incidence of immediate complications after intubation and extubation (desaturation, failure of intubation and extubation)

CONTACTS AND LOCATIONS:
Locations (1):
- Desejo Tarso Maioli, Bento Gonçalves, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nepogodiev D, Martin J, Biccard B, Makupe A, Bhangu A; National Institute for Health Research Global Health Research Unit on Global Surgery. Global burden of postoperative death. Lancet. 2019 Feb 2;393(10170):401. doi: 10.1016/S0140-6736(18)33139-8. No abstract available. PMID 30722955
- [Background] Ahmad T, Bouwman RA, Grigoras I, Aldecoa C, Hofer C, Hoeft A, Holt P, Fleisher LA, Buhre W, Pearse RM; International Surgical Outcomes Study (ISOS) group. Use of failure-to-rescue to identify international variation in postoperative care in low-, middle- and high-income countries: a 7-day cohort study of elective surgery. Br J Anaesth. 2017 Aug 1;119(2):258-266. doi: 10.1093/bja/aex185. PMID 28854536
- [Background] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Moine P, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network investigators. Incidence of mortality and morbidity related to postoperative lung injury in patients who have undergone abdominal or thoracic surgery: a systematic review and meta-analysis. Lancet Respir Med. 2014 Dec;2(12):1007-15. doi: 10.1016/S2213-2600(14)70228-0. Epub 2014 Nov 13. PMID 25466352
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Arozullah AM, Daley J, Henderson WG, Khuri SF. Multifactorial risk index for predicting postoperative respiratory failure in men after major noncardiac surgery. The National Veterans Administration Surgical Quality Improvement Program. Ann Surg. 2000 Aug;232(2):242-53. doi: 10.1097/00000658-200008000-00015. PMID 10903604
- [Background] Meara JG, Leather AJ, Hagander L, Alkire BC, Alonso N, Ameh EA, Bickler SW, Conteh L, Dare AJ, Davies J, Merisier ED, El-Halabi S, Farmer PE, Gawande A, Gillies R, Greenberg SL, Grimes CE, Gruen RL, Ismail EA, Kamara TB, Lavy C, Lundeg G, Mkandawire NC, Raykar NP, Riesel JN, Rodas E, Rose J, Roy N, Shrime MG, Sullivan R, Verguet S, Watters D, Weiser TG, Wilson IH, Yamey G, Yip W. Global Surgery 2030: evidence and solutions for achieving health, welfare, and economic development. Int J Obstet Anesth. 2016 Feb;25:75-8. doi: 10.1016/j.ijoa.2015.09.006. Epub 2015 Sep 30. No abstract available. PMID 26597405
- [Background] Wittenstein J, Ball L, Pelosi P, Gama de Abreu M. High-flow nasal cannula oxygen therapy in patients undergoing thoracic surgery: current evidence and practice. Curr Opin Anaesthesiol. 2019 Feb;32(1):44-49. doi: 10.1097/ACO.0000000000000682. PMID 30543553
- [Background] Papazian L, Corley A, Hess D, Fraser JF, Frat JP, Guitton C, Jaber S, Maggiore SM, Nava S, Rello J, Ricard JD, Stephan F, Trisolini R, Azoulay E. Use of high-flow nasal cannula oxygenation in ICU adults: a narrative review. Intensive Care Med. 2016 Sep;42(9):1336-49. doi: 10.1007/s00134-016-4277-8. Epub 2016 Mar 11. PMID 26969671
- [Background] Spence EA, Rajaleelan W, Wong J, Chung F, Wong DT. The Effectiveness of High-Flow Nasal Oxygen During the Intraoperative Period: A Systematic Review and Meta-analysis. Anesth Analg. 2020 Oct;131(4):1102-1110. doi: 10.1213/ANE.0000000000005073. PMID 32925331
- [Background] Lodenius A, Piehl J, Ostlund A, Ullman J, Jonsson Fagerlund M. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) vs. facemask breathing pre-oxygenation for rapid sequence induction in adults: a prospective randomised non-blinded clinical trial. Anaesthesia. 2018 May;73(5):564-571. doi: 10.1111/anae.14215. Epub 2018 Jan 13. PMID 29330853
- [Background] Pennisi MA, Bello G, Congedo MT, Montini L, Nachira D, Ferretti GM, Meacci E, Gualtieri E, De Pascale G, Grieco DL, Margaritora S, Antonelli M. Early nasal high-flow versus Venturi mask oxygen therapy after lung resection: a randomized trial. Crit Care. 2019 Feb 28;23(1):68. doi: 10.1186/s13054-019-2361-5. PMID 30819227
- [Background] Brainard J, Scott BK, Sullivan BL, Fernandez-Bustamante A, Piccoli JR, Gebbink MG, Bartels K. Heated humidified high-flow nasal cannula oxygen after thoracic surgery - A randomized prospective clinical pilot trial. J Crit Care. 2017 Aug;40:225-228. doi: 10.1016/j.jcrc.2017.04.023. Epub 2017 Apr 19. PMID 28454060
- [Background] Yu Y, Qian X, Liu C, Zhu C. Effect of High-Flow Nasal Cannula versus Conventional Oxygen Therapy for Patients with Thoracoscopic Lobectomy after Extubation. Can Respir J. 2017;2017:7894631. doi: 10.1155/2017/7894631. Epub 2017 Feb 19. PMID 28298878
- [Background] Fraser JF, Spooner AJ, Dunster KR, Anstey CM, Corley A. Nasal high flow oxygen therapy in patients with COPD reduces respiratory rate and tissue carbon dioxide while increasing tidal and end-expiratory lung volumes: a randomised crossover trial. Thorax. 2016 Aug;71(8):759-61. doi: 10.1136/thoraxjnl-2015-207962. Epub 2016 Mar 25. PMID 27015801
- [Background] Sklar MC, Dres M, Rittayamai N, West B, Grieco DL, Telias I, Junhasavasdikul D, Rauseo M, Pham T, Madotto F, Campbell C, Tullis E, Brochard L. High-flow nasal oxygen versus noninvasive ventilation in adult patients with cystic fibrosis: a randomized crossover physiological study. Ann Intensive Care. 2018 Sep 5;8(1):85. doi: 10.1186/s13613-018-0432-4. PMID 30187270
- [Background] Vourc'h M, Nicolet J, Volteau C, Caubert L, Chabbert C, Lepoivre T, Senage T, Roussel JC, Rozec B. High-Flow Therapy by Nasal Cannulae Versus High-Flow Face Mask in Severe Hypoxemia After Cardiac Surgery: A Single-Center Randomized Controlled Study-The HEART FLOW Study. J Cardiothorac Vasc Anesth. 2020 Jan;34(1):157-165. doi: 10.1053/j.jvca.2019.05.039. Epub 2019 May 29. PMID 31230964
- [Background] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660
- [Background] Wu X, Cao W, Zhang B, Wang S. Effect of high-flow nasal cannula oxygen therapy vs conventional oxygen therapy on adult postcardiothoracic operation: A meta-analysis. Medicine (Baltimore). 2018 Oct;97(41):e12783. doi: 10.1097/MD.0000000000012783. PMID 30313100
- [Background] Zochios V, Collier T, Blaudszun G, Butchart A, Earwaker M, Jones N, Klein AA. The effect of high-flow nasal oxygen on hospital length of stay in cardiac surgical patients at high risk for respiratory complications: a randomised controlled trial. Anaesthesia. 2018 Dec;73(12):1478-1488. doi: 10.1111/anae.14345. Epub 2018 Jul 18. PMID 30019747
- [Background] Rochwerg B, Granton D, Wang DX, Helviz Y, Einav S, Frat JP, Mekontso-Dessap A, Schreiber A, Azoulay E, Mercat A, Demoule A, Lemiale V, Pesenti A, Riviello ED, Mauri T, Mancebo J, Brochard L, Burns K. High flow nasal cannula compared with conventional oxygen therapy for acute hypoxemic respiratory failure: a systematic review and meta-analysis. Intensive Care Med. 2019 May;45(5):563-572. doi: 10.1007/s00134-019-05590-5. Epub 2019 Mar 19. PMID 30888444
- [Background] Ni YN, Luo J, Yu H, Liu D, Liang BM, Yao R, Liang ZA. Can high-flow nasal cannula reduce the rate of reintubation in adult patients after extubation? A meta-analysis. BMC Pulm Med. 2017 Nov 17;17(1):142. doi: 10.1186/s12890-017-0491-6. PMID 29149868
- [Background] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Background] Cortegiani A, Accurso G, Mercadante S, Giarratano A, Gregoretti C. High flow nasal therapy in perioperative medicine: from operating room to general ward. BMC Anesthesiol. 2018 Nov 10;18(1):166. doi: 10.1186/s12871-018-0623-4. PMID 30414608